CLINICAL TRIAL: NCT00681720
Title: An Open Label Positron Emission Tomography (PET) Study With (11C)Flumazenil to Determine Central GABAA Receptor Occupancy of AZD7325 After Oral Administration to Healthy Volunteers
Brief Title: Positron Emission Tomography (PET) Study With (11C)Flumazenil to Determine Central GABAA Receptor Occupancy of AZD7325
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, Medical Science Director, Emerging Psychiatry, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1140C00007; EudractCT 2007-005436-86
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Anxiety
Keywords: Anxiety; GABA receptors; Positron Emission Tomography; PET; phase I
MeSH Terms: conditions — Anxiety Disorders | interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide; Flumazenil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD7325; Drug: Radioligand (11C) flumazenil

INTERVENTIONS:
Drug: AZD7325 — Single dose of oral solution or capsule. 3 times per subject.
Drug: Radioligand (11C) flumazenil — Single dose of i.v solution. 4 times per subject. (3 times together with AZD7325)

SUMMARY:
The study is carried out in order to determine the relationship between the dose of AZD7325 and the blood concentration of AZD7325, and to investigate to which extent AZD7325 binds to the GABAA receptors.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18-30 kg/m2 and weight of 60-100 kg
* Clinically normal physical findings, medical history and laboratory values.

Exclusion Criteria:

* Clinically significant illness or clinical relevant trauma within 2 weeks before the study start.
* Intake of another investigational drug or participation in a clinical study the past 12 weeks.
* Previous participation in a PET study within the past 12 months. Suffer from claustrophobia and would be unable to undergo MRI (magnetic resonance imaging) or PET scanning.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography using the radioligand (11C)flumazenil | 4 times per subject

SECONDARY OUTCOMES:
To assess safety of AZD7325 by assessment of adverse events, vital signs, ECGs, physical examination, psychometric tests and laboratory variables. | 6 visits with tests for the 2 subjects in the first group (Panel 1). 7 visits with tests for the 2 subjects in the second group (Panel 2). Some tests will be done several times per visit. All tests will not be done at every visit
Investigate the pharmacokinetics of AZD7325 following single doses of AZD7325 by assessment of drug concentration in plasma | 3 times per subject. Up to 48 hours each time.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Stockholm, Sweden; Eva Taavo, Study Director — AstraZeneca R&D, Study Delivery, Clinical Development, Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden

REFERENCES:
- [Derived] Jucaite A, Cselenyi Z, Lappalainen J, McCarthy DJ, Lee CM, Nyberg S, Varnas K, Stenkrona P, Halldin C, Cross A, Farde L. GABAA receptor occupancy by subtype selective GABAAalpha2,3 modulators: PET studies in humans. Psychopharmacology (Berl). 2017 Feb;234(4):707-716. doi: 10.1007/s00213-016-4506-4. Epub 2016 Dec 24. PMID 28013354